CLINICAL TRIAL: NCT06894862
Title: A Phase I, Double-Blind, Placebo-Controlled, Randomised, First in Human, Dose Escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics of NYR-BI03 in Healthy Participants, When Administered as an Infusion for up to 6 Hours
Brief Title: A Study of the Safety, Tolerability, and Pharmacokinetics of NYR-BI03 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nyrada Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: NYR-BI03-01
Record Dates: First submitted 2025-03-09; First posted 2025-03-25 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Groups of participants are assigned to receive either NYR-BI03 or placebo in a 6:2 ratio (n=8 per cohort).
  Participants receiving the placebo will be pooled. Doses are escalated in five groups/cohorts, subject to safety review by the Safety Review Committee.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study will be conducted double blinded. Authorised unblinded study staff will be clearly designated and documented and are not permitted to perform any study assessments or have contact with participants for data collection after the first dose of study product. An unblinded pharmacist will prepare the study products and strict procedures will be implemented to ensure that only designated unblinded study staff have access to the randomized treatment allocation for each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NYR-BI03 intravenous infusion (Experimental): NYR-BI03 administered in escalating doses as a continuous intravenous infusion for up to 6 hours
  Interventions: Drug: NYR-BI03
- Placebo intravenous infusion (Placebo Comparator): Placebo comparator administered as a continuous intravenous infusion for up to 6 hours
  Interventions: Drug: Matching placebo (all cohorts)

INTERVENTIONS:
Drug: NYR-BI03 — Participants receive NYR-BI03 nanosuspension formulated for continuous intravenous infusion to be given over 3 hours or 6 hours.
  Other Names: Xolatryp
  Arms: NYR-BI03 intravenous infusion
Drug: Matching placebo (all cohorts) — Administered as a continuous intravenous infusion over 3 hours or 6 hours
  Arms: Placebo intravenous infusion

SUMMARY:
The goal of this clinical trial is to learn if investigational drug NYR-BI03 is safe and tolerated when given as an intravenous infusion for up to 6 hours to healthy male and female volunteers.

The study will also show what if any medical problems participants have when taking drug NYR-BI03 and it will provide information on blood levels of the drug.

Researchers will compare drug NYR-BI03 to a placebo (a similar substance that contains no drug) to see if NYR-BI03 is safe and tolerated.

Participants will be administered drug NYR-BI03 or a placebo via intravenous infusion for up to 6 hours and be assessed by physical examination and laboratory tests.

DETAILED DESCRIPTION:
The study is a Phase 1, double-blind, randomised, first-in-human, dose escalation study to assess the safety, tolerability, and pharmacokinetics (PK) of NYR-BI03 when administered as an intravenous (IV) infusion for up to 6 hours to healthy participants.

Six (6) ascending dose cohorts are planned. Up to 48 participants will be enrolled sequentially into the cohorts, with a total of 8 participants per cohort (6 active, 2 placebo).

Each participant will be screened within a 28-day screening period after providing voluntary, written informed consent. If eligible, participants will be admitted to the clinical unit on Day -1 for confinement and randomised to be administered a single IV dose of NYR-BI03 or placebo for up to 6 hours on Day 1.

After confinement for at least 48 hours after the start of infusion for safety assessments and collection of PK blood samples, participants will be discharged from the clinical unit on Day 3. Participants will return to the clinical unit for the End of Study visit (EOS) on Day 7 for final safety monitoring.

Safety assessments will include collection of adverse events (AEs), laboratory tests (hematology, biochemistry, coagulation, urinalysis), physical examination, basic neurological examination, pupillary response assessment, vital signs, cardiac telemetry, and 12-lead electrocardiogram (ECG). For each cohort, a sentinel group of 2 participants (1 active, 1 placebo) will be dosed at least 24 hours before the rest of the cohort.

Blinded safety and tolerability data from the sentinel group up to and including 24 hours post-dose (i.e., up to and including the Day 2 assessments) will be reviewed by the Principal Investigator, with provision for additional review if deemed necessary. Following a satisfactory safety review, dosing of the rest of the cohort may proceed.

After each completed dose cohort, the Safety Review Committee (SRC) will review the available cumulative blinded safety data and available blinded PK data.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female
* 50.0 to 105.0 kg (inclusive)
* Body Mass Index (BMI) BMI of 18.0 to 30.0 kg/m2 (inclusive)
* General Health Healthy, determined by a medical history
* Contraceptive Status: Must agree to use of established highly effective contraception for the duration of the study and for at least 30 days thereafter
* Venous Access in their left and right arm to allow collection of blood samples and drug administration.

Exclusion Criteria:

* Pregnant females and lactating females are excluded from participating in the study.
* History of allergy and/or hypersensitivity to any of the stated ingredients of the formulations.
* History of severe allergy or anaphylaxis.
* A known hypersensitivity to any surgical dressing which may be used
* History of clinically significant gastrointestinal, hepatic, renal, cardiovascular, dermatological, immunological, respiratory, endocrine, oncological, neurological, metabolic, gynecological, ear, nose, and throat, or musculoskeletal disorders, psychiatric disorder or haematological disorders
* Any history of uncontrolled, severe asthma during the last 5 years
* A creatinine clearance of less than 80 mL/min
* Any predisposing condition that might interfere with the absorption, distribution, metabolism, and/or excretion of the investigational product.
* History of abnormal bleeding tendencies, clotting disorders or thrombophlebitis unrelated to venipuncture or intravenous cannulation
* A positive test for hepatitis B surface antigen, a history of hepatitis C without a negative polymerase chain reaction (PCR) test, a history of HIV infection or demonstration of HIV antibodies
* Any evidence of organ dysfunction, or any clinically significant clinical laboratory value which, in the opinion of the Investigator would jeopardize the safety of the participant or impact on the validity of the study results,
* Liver function test (including alanine aminotransferase (ALT), aspartate aminotransferase (AST), bilirubin) or prothrombin time (PT) and activated partial thromboplastin time (aPTT) >1.5 x upper limit of normal
* Alcohol Use Those who may have difficulty abstaining from alcohol during the 48 hr prior to dose administration and until completion of the inpatient stay
* History of, or current evidence of, abuse of alcohol or any drug substance, licit or illicit, or positive urine drug screen for drugs of abuse
* Taking any prescription medications within 14 days prior to dose administration and/or likely to require prescription medication during the study
* Taking over-the-counter (OTC) medications or herbal supplements for 10 days prior to dose administration and/or likely to require or be unwilling to refrain from using OTC medications or herbal supplements during the study (with the exception of paracetamol, contraceptives, vitamin and other nutrient supplement use, at the discretion of the Investigator)
* Difficulty in abstaining from food and/or beverages that contain caffeine or other xanthines, (e.g. coffee, tea, cola and chocolate) during the 24 hr prior to dose administration and whilst confined at the clinical study facility.
* Psychiatric Disorder History of any psychiatric illness which may impair the ability to provide written informed consent
* Protocol Compliance: Poor compliers or those unlikely to attend.
* Recent Study Participation Receipt of any drug as part of a research study within 30 days or 5 half-lives, whichever is longer, of initial dose administration in this study
* Standard blood donation within the 12-week period before dose administration
* Unusual dietary habits and excessive or unusual vitamin intakes
* Vaccination or immunizations within 30 days of initial dose administration
* Participants with a risk of QT/ corrected QT interval (QTc) prolongation, namely: a. A marked baseline prolongation of corrected QTcF interval >450 ms in males and >470 ms in females in two ECGs, or b. A history of risk factors for Torsade de Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Cisgender males Cisgender females
Enrollment: 48 (Actual)
Dates: Start 2025-03-19 (Actual); Primary Completion 2025-07-24 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events | From enrollment up to and including follow-up assessments on Day 7
  The safety and tolerability of NYR-BI03 in healthy volunteers, when administered as a 3 hour or 6 hour intravenous (IV) infusion.

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of NYR-BI03 | For 3-hour infusion: Pre-infusion, +10minutes, +30 minutes, 1, 2, 3, 3.5, 4, 6 , 9 hours. For 6-hour infusion: Pre-infusion, +10minutes, +30 minutes and 1, 3, 4, 6, 6.5, 7, 9, 12, 24 hours.
  Blood samples taken at regular intervals pre and post the start of infusion
Maximum observed blood concentration (Cmax) of NYR-BI03 | For 3-hour infusion: Pre-infusion, +10minutes, +30 minutes, 1, 2, 3, 3.5, 4, 6 , 9 hours. For 6-hour infusion: Pre-infusion, +10minutes, +30 minutes and 1, 3, 4, 6, 6.5, 7, 9, 12, 24 hours.
  Blood samples taken at regular intervals pre and post the start of infusion
Tmax (time of occurrence of Cmax) of NYR-BI03 | For 3-hour infusion: Pre-infusion, +10minutes, +30 minutes, 1, 2, 3, 3.5, 4, 6 , 9 hours. For 6-hour infusion: Pre-infusion, +10minutes, +30 minutes and 1, 3, 4, 6, 6.5, 7, 9, 12, 24 hours.
  Blood samples taken at regular intervals pre and post the start of infusion
Apparent terminal half-life (T1/2) of NYR-BI03 | For 3-hour infusion: Pre-infusion, +10minutes, +30 minutes, 1, 2, 3, 3.5, 4, 6 , 9 hours. For 6-hour infusion: Pre-infusion, +10minutes, +30 minutes and 1, 3, 4, 6, 6.5, 7, 9, 12, 24 hours.
  Blood samples taken at regular intervals pre and post the start of infusion
Total body clearance from blood (CL) of NYR-BI03 calculated as Dose/AUC | For 3-hour infusion: Pre-infusion, +10minutes, +30 minutes, 1, 2, 3, 3.5, 4, 6 , 9 hours. For 6-hour infusion: Pre-infusion, +10minutes, +30 minutes and 1, 3, 4, 6, 6.5, 7, 9, 12, 24 hours.
  Blood samples taken at regular intervals pre and post the start of infusion

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Argent, MD, Principal Investigator — Scientia Clinical Research Ltd
Locations (1):
- Scientia Clinical Research Ltd, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified individual participant data along with key supporting documents (protocol, statistical analysis plan, data dictionary, clinical study report, and case report forms).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available 12 months after publication of primary results and remain accessible for at least 5 years.
Access Criteria: Data access requests will be evaluated by an independent Data Access Committee. Applicants must submit a research proposal and evidence of ethics approval, and, if approved, sign a data use agreement that restricts use to the proposed research and prohibits re-identification. Data will be hosted in a secure repository. For inquiries, please contact Dr Alexandra Suchowerska at alexandra.suchowerska@nyrada.com